CLINICAL TRIAL: NCT03800914
Title: High Intensity Interval Training in Fibrotic Interstitial Lung Disease: a Randomized Controlled Trial
Brief Title: High Intensity Interval Training in Fibrotic Interstitial Lung Disease
Acronym: HIIT in fILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Anne E Holland PhD, FThorSoc, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LTU HIIT in ILD
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Fibrotic Interstitial Lung Disease
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Interval Training (Experimental): Participants will undergo a twice-weekly supervised exercise training program for eight weeks. Each session will involve 36 minutes of interval aerobic exercise on a cycle ergometer alternating every 30 seconds between 100% of peak work rate, achieved on the cardiopulmonary exercise test (CPET), plus upper and lower resistance training.
  Interventions: Other: High intensity interval training
- Traditional pulmonary rehabilitation (Active Comparator): Participants will undergo a twice-weekly supervised exercise training program for eight weeks. Each session will involve 30 minutes of continuous aerobic exercise on a cycle ergometer at 60% of the peak work rate achieved on the CPET, plus upper and lower resistance training.
  Interventions: Other: Traditional pulmonary rehabilitation

INTERVENTIONS:
Other: High intensity interval training — 36 minutes of interval exercise on cycle ergometer alternating every 30 seconds between 100% peak work rate achieved on cardiopulmonary exercise test and unloaded cycling
  Arms: High Intensity Interval Training
Other: Traditional pulmonary rehabilitation — 30 minutes of continuous exercise on cycle ergometer at 60% peak work rate achieved on cardiopulmonary exercise test.
  Arms: Traditional pulmonary rehabilitation

SUMMARY:
The fibrotic interstitial lung diseases (fILD) is a group of debilitating chronic lung conditions that are characterised by scarring of lung tissue, dyspnoea on exertion and significant physical impairment. Exercise training is recommended for people with fILD in improving breathlessness and exercise tolerance. However, despite the best efforts of patients and clinicians, many of those who participate are not attaining its benefits. The current exercise training strategies of moderate intensity continuous training may not be well suited to fILD. High intensity interval training (HIIT), short bouts of high-intensity exercise regularly interspersed with periods of rest or light exercise may be an alternate exercise training option for people with fILD.

The study will determine to whether HIIT is better than the current method of continuous exercise training at moderate intensity in improving exercise tolerance, breathlessness and quality of life in people with fILD. A randomised controlled, assessor blinded trial will be conducted. A total 130 people with fILD will be randomly assigned to moderate intensity continuous training or HIIT. If this trial demonstrates that HIIT is effective, it will provide an exercise training strategy that can readily be implemented in practice that will maximise the outcomes of exercise training for people with fILD.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a chronic lung condition characterized by scarring of lung tissue. This stiffening of the lungs impairs breathing and reduces the amount of oxygen being delivered throughout the body limiting the ability to perform daily and physical activity. Around two-thirds of people with ILD have fibrotic ILD (fILD), a type of ILD, which typically has worse impairment and disability than other types of ILD. There is no cure for these conditions, although there are two new pharmacological therapies that slow the decline in lung function in Idiopathic Pulmonary Fibrosis (IPF), the most common type of fILD. These treatments however do not provide improvement in breathlessness, exercise capacity or health-related quality of life (HRQoL).

Exercise training, or Pulmonary Rehabilitation (PR), has shown to be effective at improving exercise tolerance and HRQoL in ILD. The investigators recently demonstrated that, at a group level, exercise training exerts a positive effect across varying subtypes of ILD, including IPF, the most rapidly progressive of all the fILDs. However less than half of those with IPF who undertook the exercise training achieved meaningful improvements in exercise capacity. In addition, a large proportion of people with IPF were unable to keep up with the recommended exercise training level, often due to excessive dyspnoea or desaturation. This suggests the current exercise training strategies used in PR, which were adopted from guidelines for patients with chronic obstructive pulmonary disease (COPD), may not provide the optimal exercise stimuli for fILD. High intensity interval training (HIIT), which is short bouts of high intensity exercise regularly interspersed with periods of rest or light exercise, may be an alternate exercise training option for people with fILD. However, it is unknown whether this kind of exercise training achieves superior benefits to the traditional model of PR.

The aim of this project is to determine whether HIIT is better than the current method of continuous exercise training at moderate intensity, in improving exercise capacity, breathlessness and HRQoL in people with fILD. A total 130 people with fILD will be recruited. The trial will be conducted at four hospital sites across Australia. People who agree to take part in the study will be randomly allocated into two groups. Group 1 will undergo the traditional PR model of moderate intensity continuous exercise training and group 2 will undergo HIIT. Participants in both groups will participate in exercise training twice weekly for eight weeks. The participants will be monitored continuously during exercise by an experienced physiotherapist or exercise physiologist. At the beginning and the end of the eight weeks of exercise training, and six months later, participants will undergo measurements of exercise capacity and health status. This study will determine whether HIIT is effective, providing an important exercise training strategy that can be readily used for people with fILD to achieve positive benefits from PR.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibrotic interstitial lung disease (fILD)
* Able to read and speak English

Exclusion Criteria:

* Resting oxygen saturation (SpO2) is < 85%
* Severe pulmonary hypertension (WHO class IV)
* Attendance at Pulmonary rehabilitation (PR) within last 12 months
* Comorbidities which preclude exercise training
* History of syncope on exertion
* Significant cognitive impairment
* Anticipated transplant or death within the duration of the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in endurance time | Baseline, nine weeks and 6 months following intervention
  Endurance time measured during constant work rate test (CWRT) at 75% of the peak work rate achieved on a baseline cardiopulmonary exercise test (CPET).

SECONDARY OUTCOMES:
Change in dyspnea measured using the Dyspnea-12 questionnaire | Baseline, nine weeks and 6 months following intervention
  Dyspnea-12 is a uni-dimensional 12-item questionnaire divided in 2 domains: physical items (1 to 7) and affective items (8-12). Each item evaluate breathing experience and can be scored as: None (0), Mild (1), Moderate (2) or Severe (3). Results of this questionnaire will be reported as total score that can range from 0 to 36 and separate scores that can range from 0 to 21 for physical component and 0 to 15 for affective component. Higher scores indicate worse dyspnea.
Changes in fatigue evaluated by the Fatigue Severity Scale | Baseline, nine weeks and 6 months following intervention
  Fatigue Severity Scale (FSS), a self reported rating scale including 9 items to measure how fatigue affects motivation, exercise, physical functioning, carrying out duties and how fatigue interferes with work, family, or social life. Each item is scored on a 7 point scale in which 1 = strongly disagree and 7= strongly agree. Total score range from 9 to 63. Higher scores indicate greater fatigue severity.
Change in health related quality of life using the St George's Respiratory Questionnaire idiopathic pulmonary fibrosis specific version (SGRQ-I) | Baseline, nine weeks and 6 months following intervention
  The SGRQ-I is a disease specific HRQoL measure with similar psychometric properties to the original SGRQ that is designed to be more relevant in patients with IPF. The questionnaire is divided in 3 domains: Symptoms (frequency and severity), Activity (activities that cause or are limited by breathlessness) and Impact (social functioning and psychological disturbances resulting from airways disease). Values of each domain as well as the total score value will be reported. Each item is weighted based on empirical data. Total score and scores in each domain can range from 0 to 100. Higher scores indicate more limitations in quality of life.
Change in health related quality of life using the chronic respiratory disease questionnaire (CRQ) | Baseline, nine weeks and 6 months following intervention
  The CRQ consists of 20 items across 4 domains: Dyspnea (activities that cause breathlessness and are performed frequently), fatigue, emotional function and mastery ( the patient's feeling of control over their disease). Each domain includes four to seven items, and each item is scored on a 7-point Likert score. Total scores for each domain range from 4-35. Values of each domain will be reported. Lower scores indicate more limitations in quality of life.
Change in anxiety and depression measured by the Hospital Anxiety and Depression Scale | Baseline, nine weeks and 6 months following intervention
  Hospital Anxiety and Depression Scale (HADS), a scale with 14 items divided into two domains : anxiety symptoms (7 items) and depression symptoms (7 items). Each item can be scored from 0 to 3. Scores from each domain can vary from 0 to 21 and are stratified as follows: 0-7 (indicates absence of anxiety/depression symptoms); 8-10 ( presence of symptoms of anxiety and depression in moderate degree - borderline); 11 or more (significant number of anxiety/depression symptoms - confirmed cases). Score of each domain as well as number of confirmed cases will be reported.
Change in functional exercise capacity assessed by 6-minute walk distance | Baseline, nine weeks and 6 months following intervention
  Distance in meters achieved on a 6-minute walk test
Changes in skeletal muscle size | Baseline, nine weeks and 6 months following intervention
  Change in cross-sectional area of the Quadriceps will be measured by B-mode ultrasonography
Dyspnea related disability - measured with modified medical research council scale (MMRC) | Baseline, nine weeks and 6 months following intervention
  The MMRC rates dyspnea according to different levels activity on a 5-point scale (grade 0-4), with grade 4 representing the greatest level of dyspnea impairment.
Global rating of change | Baseline, nine weeks and 6 months following intervention
  The global rating of change will assess the participants' overall self-perceived change in health by asking the participant to rate their change as either 'worse', 'about the same' or 'better'. The extent of change ( (i.e., worsening or improvement) is then graded on a Likert scale from one to seven.
Change in physical activity | Baseline, nine weeks and 6 months following intervention
  Time spent sedentary and in physical activity of various intensities will be measured by a wrist-worn, tri-axial accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holland, Study Director — Monash University
Locations (4):
- Australia (4):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Prince Charles Hospital, Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowman LM, May AK, Hill CJ, Bondarenko J, Spencer L, Morris NR, Alison JA, Walsh J, Goh NSL, Corte T, Glaspole I, Chambers DC, McDonald CF, Holland AE. High intensity interval training versus moderate intensity continuous training for people with interstitial lung disease: protocol for a randomised controlled trial. BMC Pulm Med. 2021 Nov 10;21(1):361. doi: 10.1186/s12890-021-01704-2. PMID 34758808